CLINICAL TRIAL: NCT01736605
Title: The Effect of Meditation and Massage Therapy for Breast Cancer Patients Undergoing Autologous Tissue Reconstruction - A Pilot Study
Brief Title: The Effect of Meditation and Massage Therapy for Breast Cancer Patients Undergoing Tissue Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dietlind Wahner-Roedler, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-008563
Record Dates: First submitted 2012-11-20; First posted 2012-11-29 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Breast Cancer
Keywords: Massage; Meditation; Breast Cancer; Breast Surgery; Breast Reconstruction
MeSH Terms: conditions — Breast Neoplasms | interventions — Massage; Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Massage (Active Comparator): Daily massage for 20 minutes the first 3 days following surgery.
  Interventions: Procedure: Massage
- Massage combined with meditation (Active Comparator): Daily massage for 20 minutes combined with meditation the first 3 days following surgery.
  Interventions: Procedure: Massage combined with meditation

INTERVENTIONS:
Procedure: Massage — Patients will receive a daily 20 minute massage in their hospital room on the first 3 days following surgery.
  Arms: Massage
Procedure: Massage combined with meditation — Patients will receive a daily 20 minute massage combined with meditation in their hospital room on the first 3 days following surgery.
  Other Names: Massage; Meditation
  Arms: Massage combined with meditation

SUMMARY:
In this study we propose to explore the efficacy of massage therapy combined with meditation in women recovering from tissue reconstruction after mastectomy for breast cancer. Patients will be randomized into 2 groups. The first group will consist of massage therapy on 3 consecutive days starting on the 1st day after surgery. The second group will consist of massage therapy combined with meditation for 3 consecutive days starting on the 1st day after surgery. The effect of massage and massage combined with meditation on stress, anxiety, relaxation, insomnia, alertness, fatigue, tension/muscular discomfort, pain, mood and energy level will be evaluated by using three different surveys.

DETAILED DESCRIPTION:
Besides skin cancer breast cancer is the most common malignancy among women. Most women with breast cancer will undergo some kind of breast cancer surgery. For women undergoing a mastectomy, breast reconstruction offers significant quality of life benefits and is a vital option to enhance breast cancer recovery. There are two general types of reconstructive options:

1. Prosthetic devices (saline implants, silicone implants, tissue expanders)
2. Autologous tissue reconstructions with tissue flaps that are transferred from adjoining or distant donor sites to the anterior chest wall.

When reconstruction of the breast mound is accomplished using the patient's own tissues, the result is typically more natural in both appearance and feel than with expander/implant reconstruction. However the disadvantages of autologous reconstruction include longer surgical procedures and prolonged recovery time as compared to prosthetic reconstruction. Postoperative pain, anxiety, fatigue are among the challenges facing patients undergoing breast cancer surgery and especially patients who decided to undergo these complicated plastic surgical procedures. Massage therapy has been used successfully to target common postoperative symptoms such as pain, anxiety, tension and fatigue in breast cancer patients.

Meditation has been shown to be helpful in achieving healing and relaxation through purposeful contemplation and reflection.

In this study we propose to explore the effectiveness of massage therapy combined with meditation in breast cancer patients recovering from autologous tissue reconstruction with the hope that the combination will augment the benefit obtained by massage therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 and above able to give informed consent
* Women who are undergoing mastectomies for breast cancer and the following autologous tissue reconstruction.

  * Free TRAM flaps (TRAM = Transverse Rectus Abdominis Myocutaneous)
  * Muscle-sparing (MS) free TRAM flaps (or MS-TRAM)
  * DIEP flaps (DIEP = Deep Inferior Epigastric Perforator)
  * SIEA flaps (SIEA = Superficial Inferior Epigastric Artery)
  * Pedicled TRAM flaps
* Patients who undergo one of these 5 surgeries on a Monday or a Tuesday
* Able to speak and understand English
* Able to complete the three questionnaires

Exclusion Criteria:

* Women who decline to participate in the study
* Women with any kind of breast reconstruction surgery other than what is listed in the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Assess the effect of massage therapy on pain and stress related symptoms after breast reconstruction surgery compared to baseline. | 3 Days

SECONDARY OUTCOMES:
Assess the effect of massage therapy combined with meditation on pain and stress related symptoms after breast reconstruction surgery compared to baseline. | 3 Days

CONTACTS AND LOCATIONS:
Overall Officials: Dietlind L. Wahner-Roedler, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States